CLINICAL TRIAL: NCT05515224
Title: 5-Cog Paradigm to Improve Detection of Cognitive Impairment in Primary Care: Pragmatic Clinical Trial
Brief Title: 5-Cog 2.0: A Pragmatic Clinical Trial
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Albert Einstein College of Medicine (Other)
Collaborators: Indiana University (Other); National Institute of Neurological Disorders and Stroke (NINDS) (NIH); Northwestern University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: 2022-14144; 2U01NS105565-07 (NIH)
Record Dates: First submitted 2022-08-23; First posted 2022-08-25 (Actual); Last update posted 2025-03-17 (Actual); Status verified 2025-03

CONDITIONS: Dementia; Cognitive Impairment
MeSH Terms: conditions — Dementia; Cognitive Dysfunction

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 5-Cog Paradigm (5-Cog battery coupled with clinical decision tool) (Experimental): A cognitive concern screening will be conducted with patients aged 65 and older prior to their appointment with their primary care physician. If cognitive concerns are endorsed the 5-Cog battery will be conducted. The simple, <5-minute cognitive assessment will reliably identify older persons with cognitive impairment in primary care settings, and flag them for further evaluation. Depending on whether the 5-Cog results are normal or abnormal on any one of the 3 tests, appropriate clinical decision support tools are provided to the primary care physicians in electronic medical record. The primary care physicians are not instructed to follow 5-Cog suggestions verbatim but use their clinical judgment.
  Interventions: Other: 5-Cog Paradigm (5-Cog battery coupled with clinical decision tool)
- Enhanced usual care (Active Comparator): Educational sessions for primary care physicians and clinic staff regarding cognitive detection and medical billing will be conducted. A cognitive concern screening will be conducted with patients aged 65 and older prior to their appointment with their primary care physician. The results will be provided to primary care physicians.
  Interventions: Other: Enhanced usual care

INTERVENTIONS:
Other: 5-Cog Paradigm (5-Cog battery coupled with clinical decision tool) — A cognitive concern screening will be conducted with patients aged 65 and older prior to their appointment with their primary care physician. If cognitive concerns are endorsed the 5-Cog battery will be conducted. The 5-Cog battery includes the Picture Memory Impairment Screen, Motoric Cognitive Risk Syndrome diagnosis, and Symbol Match. The simple, <5-minute cognitive assessment will reliably identify older persons with cognitive impairment in primary care settings, and flag them for further evaluation.
  Arms: 5-Cog Paradigm (5-Cog battery coupled with clinical decision tool)
Other: Enhanced usual care — A cognitive concern screening will be conducted with patients aged 65 and older prior to their appointment with their primary care physician. The results will be provided to primary care physicians.
  Arms: Enhanced usual care

SUMMARY:
Cognitive impairment related to dementia is frequently under-diagnosed in primary care settings. This problem is more prevalent in health disparities populations. The investigators developed the 5-Cog brief cognitive assessment that is simple to use, standardized, takes <5 minutes, does not require informants, and accounts for major technical, cultural, and logistical barriers of current assessments. The investigators propose a hybrid Type 1 effectiveness-implementation design in real-world settings to adapt and test the effectiveness of the 5-Cog paradigm to increase detection of cognitive impairment care in older adults presenting with cognitive concerns.

The study aim is to evaluate, using a pragmatic cluster-randomized trial design, the effectiveness of the 5-Cog paradigm to increase 'incident cognitive impairment' detection (new MCI and dementia diagnoses) relative to enhanced usual care in 6,600 older patients presenting with cognitive concerns in 22 primary care clinics in Bronx and Indiana. As diagnosis without action will not improve patient care, 'improved dementia care' will be examined as a secondary outcome. Results will also be examined in NIH designated health disparity populations including underserved minority and socio-economically challenged populations.

DETAILED DESCRIPTION:
Cognitive impairment related to dementia is frequently under-diagnosed in primary care settings despite the increasing rates of patient cognitive complaints and the availability of numerous cognitive assessment tools. Missed detection delays treatment of reversible conditions as well as provision of support services and critical planning. This problem is more prevalent among older African-Americans and Hispanics than older whites, and more common in rural than urban populations.

The investigators developed the 5-Cog brief cognitive assessment that is simple to use, standardized, takes <5 minutes, does not require informants, and accounts for major technical, cultural, and logistical barriers of current assessments. The investigators are conducting a simple randomized clinical trial to examine the clinical efficacy of the 5-Cog paradigm (5-Cog brief cognitive assessment paired with a clinical decision-making tool) to improve dementia care in 1,200 predominantly minority sample of older adults with cognitive concerns presenting to a primary care clinic in the Bronx. Interim analysis revealed that the 5-Cog paradigm resulted in an over 8-fold increase in new cognitive impairment diagnoses and over 3-fold increase in improved dementia care actions by primary care physicians compared to an active control arm. Following up on these very promising results, the investigators propose a hybrid Type 1 effectiveness-implementation design in real-world settings to adapt and test the effectiveness of the 5-Cog paradigm to increase detection of cognitive impairment care in older adults presenting with cognitive concerns.

The aim of the pragmatic cluster-randomized trial is to test the clinical effectiveness of the 5-Cog paradigm in increasing cognitive impairment detection and improving dementia care - ascertained via electronic medical record. Randomization will be at the clinic level, and select 22 primary care practices; 6 in Bronx and 18 in urban and rural Indiana. 300 participants per practice will be enrolled for a total of 6,600 older patients with cognitive concerns. Results will also be examined in NIH designated health disparity populations including underserved minority and socio-economically challenged populations.

Outcomes are new cognitive impairment diagnoses (primary) and improved dementia care (secondary) in the 90-day period following presentation of cognitive concern to the primary care physician.

* New cognitive impairment diagnoses (primary): New diagnosis of dementia or Mild Cognitive Impairment by primary care physicians. For patients with a previous diagnosis of Mild Cognitive Impairment in electronic medical record, only a new diagnosis of dementia will be considered as an incident outcome.
* Improved dementia care (secondary): Any of the following: 1. Tests ordered for reversible causes of cognitive impairment as per published guidelines. 2. New cognitive enhancing medication prescriptions or deprescribing anti-cholinergic. 3. Referral for cognitive/dementia evaluation by specialists (Neurology, Geriatrics, Psychiatry). 4. Referral to social worker or community-based organizations.

Implementation issues and cost-effectiveness of the 5-Cog paradigm will also be examined.

This proposed study focuses on scalable approaches to address the unmet need of early detection of incident cognitive impairment, including in populations that experience health disparities.

ELIGIBILITY:
Inclusion Criteria:

1. 65 years and older
2. Presence of cognitive concerns
3. English or Spanish speaking.
4. Able to see and hear well enough to complete assessments.

Exclusion Criteria:

1. Prior diagnosis of dementia (documented in the electronic medical record or reported by physicians).
2. Permanent nursing facility residents.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 6600 (Estimated)
Dates: Start 2023-08-18 (Actual); Primary Completion 2027-11 (Estimated); Study Completion 2027-11 (Estimated)

PRIMARY OUTCOMES:
New cognitive impairment diagnoses in the 90-day period following presentation of cognitive concern to the primary care physician (PCP). | 90 days
  The clinical effectiveness of the 5-Cog paradigm on new cognitive impairment detection will be examined by comparing the proportion of 'new Mild Cognitive Impairment (MCI) and dementia diagnoses' over 90-days in the 5-cog paradigm and the enhanced usual care group using generalized linear mixed effects models. For patients with a previous diagnosis of MCI in the electronic medical record, only a new diagnosis of dementia will be considered as an incident outcome.

SECONDARY OUTCOMES:
Improved dementia care in the 90-day period following presentation of cognitive concern to the primary care provider (PCP). | 90 days
  The clinical effectiveness of the 5-Cog paradigm on improved dementia care will be examined by comparing the proportion of documentation of improved dementia care in the 5-cog paradigm and the enhanced usual care group using generalized linear mixed effects models. Improved dementia care is defined as any of the following: 1. Tests ordered for reversible causes of cognitive impairment as per published guidelines. 2. New cognitive enhancing medication prescriptions or deprescribing anti-cholinergic. 3. Referral for cognitive/dementia evaluation by specialists (Neurology, Geriatrics, Psychiatry). 4. Referral to social worker or community-based organizations.

CONTACTS AND LOCATIONS:
Overall Officials: Joe Verghese, MD, Principal Investigator — Stony Brook University; Malaz Boustani, MD, MPH, Principal Investigator — Indiana University; Erica Weiss, PhD, Principal Investigator — Albert Einstein College of Medicie
Locations (2):
- United States (2):
  - Indiana University, Bloomington, Indiana
  - Albert Einstein College of Medicine, The Bronx, New York

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data for all primary and secondary outcome measures will be made available with appropriate ethics committee and data sharing agreements in place.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will be available within 1 year of study completion.
Access Criteria: Data access requests will be reviewed by the PI and Steering Committee. Requestors will be required to sign a Data Access Agreement.

REFERENCES:
- [Derived] Chalmer RBR, Ayers E, Weiss EF, Fowler NR, Telzak A, Summanwar D, Zwerling J, Wang C, Xu H, Holden RJ, Fiori K, French DD, Nsubayi C, Ansari A, Dexter P, Higbie A, Yadav P, Walker JM, Congivaram H, Adhikari D, Melecio-Vazquez M, Boustani M, Verghese J. Improving Early Dementia Detection Among Diverse Older Adults With Cognitive Concerns With the 5-Cog Paradigm: Protocol for a Hybrid Effectiveness-Implementation Clinical Trial. JMIR Res Protoc. 2025 Apr 3;14:e60471. doi: 10.2196/60471. PMID 40179383